CLINICAL TRIAL: NCT07310290
Title: PHASES: Prodrome in tHe reAl World: aSsESsing Ubrogepant Acute Use
Brief Title: Study to Assess the Real-World Effectiveness of Ubrogepant in Adult Participants When Treating During the Prodrome Phase of Migraine Attacks
Acronym: PHASES
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-590
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Migraine; Ubrogepant; UBRELVY
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ubrogepant: Participants will receive Ubrogepant as prescribed by their physician according to local label.

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headaches, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will assess changes in migraine attack severity for adult participants treating with oral ubrogepant across migraine attacks.

Ubrogepant is a drug that is approved for the acute treatment of migraine in adults. Approximately 189 participants will be enrolled in approximately 15 sites across the US.

Participants will receive ubrogepant as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 13 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* History of 4 to 10 migraine days per month with moderate to severe headache pain in each month of the 3 months prior to Visit 1

  --a. Participants with a diagnosis of chronic migraine who report having 4 to 10 migraine days per month with moderate to severe headache pain in each month of the 3 months prior to Visit 1 due to concomitant preventive treatment are allowed in the study
* Participant is currently prescribed ubrogepant and has been using ubrogepant for at least 3 months for the acute treatment of migraine in adults, according to the US Food and Drug Administration (FDA)-approved indication
* Adult participants with current clinical diagnosis of migraine or chronic migraine according to International Classification of Headache Disorders (ICHD)-3

Exclusion Criteria:

* Currently participating in a concurrent clinical or non-interventional study.
* Concomitant use with a strong Cytochrome P450 3A4 (CYP3A4 ) inhibitor.
* Current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia, status migrainosus or painful cranial neuropathy as defined by ICHD-3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants receiving ubrogepant per routine clinical care for the treatment of migraine in the US.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Absence of moderate to severe headache over 24 hours post-dose during prodrome. | Up to approximately 13 weeks
  Prodrome is often the earliest phase of migraine attack and consists of various symptoms including sensitivity to light, fatigue, neck pain, sensitivity to sound, dizziness and difficulty thinking/concentrating.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Neurology and Pain Specialty Center /ID# 278508, Aliso Viejo, California
  - Chicago Headache Center & Research Inst /ID# 272345, Naperville, Illinois
  - Tri City Research Center, LLC /ID# 278800, Grand Island, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-590